CLINICAL TRIAL: NCT02827214
Title: Thoracolumbar Burst Fractures (AOSpine A3, A4) in Neurologically Intact Patients: An Observational, Multicenter Cohort Study Comparing Surgical Versus Non-surgical Treatment
Brief Title: Thoracolumbar Burst Fractures Study Comparing Surgical Versus Non-surgical Treatment
Status: Completed | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Collaborators: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Other Study IDs: Spine_TL-A3-A4
Record Dates: First submitted 2016-05-23; First posted 2016-07-11 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Thoracolumbar Burst Fracture
Keywords: Thoracolumbar spine; Burst fractures; Conservative treatment; Surgical treatment; Thoracic or lumbar vertebrae

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical treatment: Several surgical treatments exist to treat the fractures included in the study. The following section describes the different surgical treatment modalities in more detail
  Approaches:
  * Open short segment surgical fixation (1 level above and below the fracture level) with or without posterior decompression
  * Open long segment posterior fixation (2 or more levels above, 2 or more levels below) with or without posterior decompression
  * Posterior short or long fixation with posterolateral corpectomy and reconstruction
  * Anterior alone instrumentation
  * Combined Anterior Posterior (AP) instrumentation
  * Percutaneous posterior fixation combined with anterior instrumentation
  * Percutaneous posterior fixation with or without vertebroplasty
- Non-surgical treatment: Non-surgical treatment is defined as bed rest followed by immobilization with:
  * Custom-molded or prefabricated total body contact thoracolumbosacral orthosis (TLSO)
  * Thermoplastic removable brace
  * Jewett hyperextension braces
  * Anterior hyperextension brace (ASH)
  * Taylor-Knight brace
  * Plaster of Paris (POP)

SUMMARY:
Thoracolumbar (TL) burst fractures in neurologically intact patients account for approximately 45% of all TL spine injuries. Despite being common fractures, there is significant variability in treatment recommendations encompassing surgery and non-surgical treatment options. The controversy regarding optimal treatment for these injuries is fueled by several studies which suggest a potential benefit to surgical treatment in the realm of patient satisfaction, and the overall socio-economic burden of treatment while other studies demonstrate improved outcomes and lower morbidity with non-surgical treatment. This study aims to perform a prospective cohort analysis investigating the clinical outcome of various treatment alternatives for patients with A3/A4 fractures in the thoracolumbar region. A cost-effectiveness analysis will also be performed to identify costs and benefits of each treatment option. More specifically a sub-group analysis will be performed for this group of patients, which have equipoise in regards to patients treatment, as decided by a blinded review panel.

DETAILED DESCRIPTION:
208 subjects (i.e., 137 per surgical group; 71 per conservative group) with TL burst fractures AOSpine classification type A3 or A4 without neurological deficit as defined in the inclusion/exclusion criteria, and with or without suspected Posterior Ligament Complex (PLC) injury (M1) from T10 to L2, will be enrolled in a prospective multicenter cohort study. Patients may have an associated B injury, but must have an A3 or A4. Patients will be monitored prospectively for patient reported, clinical and radiologic outcomes, over a period of 2 years post-treatment. Specifically a patient diary will measure the Oswestry Disability Index (ODI), and employment information (indirect costs questionnaire) every second week until 6 months post-treatment. Diary will continue every second month until 2 years post-treatment. All interventions/examinations are considered as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature, age 18 to 65 years old inclusive
* Diagnosis of AO type A3 or A4 fractures on a CT scan with or without a suspected PLC injury (M1) from T10 to L2.
* Patients may have an associated B injury, but must have an A3 or A4.
* TLICS Score between 2-5 inclusive
* Acute fracture - diagnosis and treatment within 10 days of injury
* Ability to understand the content of the patient information / informed consent form
* Willingness and ability to participate in the clinical investigation including imaging and FU procedures
* Investigation according to the Clinical Investigation Plan (CIP)
* Signed and dated IRB/EC-approved written informed consent

Exclusion Criteria:

* Any neurological deficit associated with the fracture. Absence of neurological deficit will be determined with the International Standards for Neurological Classification of Spinal Cord Injury (ISNC SCI). It will be documented the status "E" (neurologically intact/normal) of the patient.
* Spontaneous fractures due to pathologic processes or neoplasia
* Head injuries causing inability to cooperate during hospital admission
* Open or penetrating spinal lesion (e.g. due to gun, stab, or projectile)
* Prior spinal surgeries in thoracic or lumbar spine
* Additional musculoskeletal, head or other injuries which would preclude rapid mobilization
* Multiple trauma or Injury Severity Score (ISS) > 16
* Other co-morbidities precluding the patient to be considered as a surgical or non-surgical candidate, i.e. burns, dementia, BMI > 40, etc.
* Any severe systemic medical disease that would exclude the patient to be a potential candidate for surgery
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study
* Recent history of substance abuse (i.e., recreational drugs, alcohol) that would preclude reliable assessment.
* Pregnancy or women planning to conceive within the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thoracolumbar burst fractures
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 1 year
  ODI within the first year after surgical or non-surgical treatment using time to event analysis

SECONDARY OUTCOMES:
AOSpine Patient Reported Outcome Spine Trauma (AOSpine Prost) | 2 years
  AOSpine PROST consists of 19 questions on aspects of functioning such as personal care, traveling, and emotional functioning after the accident causing the spinal injury. Each item has a 0-100 numeric rating scale, supported by smileys at both ends of the ruler. It is important to realize that 0 indicates a level at which the patient is non-functional and 100 indicates the level before the accident, no matter how well or poorly the patient functioned before the accident.
Quality of life EQ5D-3L | 2 years
  The EuroQoL-5D (EQ-5D) is a standardized instrument that was designed for self-completion. It has five items (mobility, self-care, usual activities, pain / discomfort and anxiety / depression) with a three-point categorical response scale (1 = no problems, 2 = some / moderate problems, 3 = extreme problems) where the patient's current health status will be assessed.
Numeric Pain Rating Scale (NPRS) | 2 years
  The NPRS measures the subjective intensity of pain. The patient is asked to make a pain rating, corresponding to his/her experienced pain.
Spine Adverse Events Severity System (SAVES) | 2 years
  The SAVES is a prospective adverse event (AE) recording instrument. The AEs are defined as any unexpected or undesirable events occurring as a result of spinal surgery, and a complication as a disease or disorder, which, as a consequence of a surgical procedure, that will negatively affect the outcome of a patient.
overall satisfaction with the treatment | 2 years
  The overall satisfaction with treatment questionnaire contents one question regarding the satisfaction with the results of the recent treatment of the spine injury with a rating system from extremely satisfied (1) to not sure/no opinion (8)
Non-surgical treatment failure rate | 2 years
  Failure rate of conservative treatment will be assessed during this study. Non-surgical treatment failure is defined as necessity of surgery after non-surgical treatment.
Surgical treatment failure rate | 2 years
  Surgical treatment failure is defined as necessity of an additional surgery after the primary surgical treatment.
indirect cost questionnaire | 2 years
  The indirect cost questionnaire assesses the personal situation of the patient at his workplace regarding to health, support, and their financial income statement
Validation of AO TL Classification System aided by the analysis of CT scans | 2 years
  The participating clinics will upload the clinical data (de-identified X-rays, CT, MRI images) on a secure web-based platform. AOSpine Knowledge Forum Trauma Steering committee members, blinded to the diagnosis made in the study, will analyze the different images to validate the different TL fractures type A3 or A4 with or without PLC injury according to the new AOSpine TL Classification System.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Dvorak, MD, Principal Investigator — Vancouver General Hospital
Locations (14):
- United States (4):
  - University of California, San Diego Medical Center, San Diego, California
  - SUNY Upstate, East Syracuse, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - West Virginia University, Morgantown, West Virginia
- Alfred Health operating through the Alfred hospital, Melbourne, Australia
- Canada (2):
  - Hopital l'Enfant-Jesus, CHU de Quebec, Québec
  - Vancouver General Hospital, Vancouver
- Assiut University Hospitals, Asyut, Egypt
- KAT Hospital, Kifissia, Greece
- Ganga Hospital, Coimbatore, India
- UMC Utrecht, Utrecht, Netherlands
- Clinical Hospital "Prof. N.Oblu", Iași, Romania
- Hospital Universitario Costa del Sol, Marbella, Spain
- Inselspital, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's website — https://www.aofoundation.org